CLINICAL TRIAL: NCT02436746
Title: The Cognitive Variability in Neurofibromatosis Type I and Tuberous Sclerosis Complex Monozygotic Twins
Brief Title: The Cognitive Variability in NF1 and TSC Monozygotic Twins
Acronym: COVANTT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, M.C.Y. de Wit, MD PhD, Prof. Y. Elgersma, Erasmus Medical Center
Other Study IDs: MEC-2014-483
Record Dates: First submitted 2015-04-29; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Neurofibromatosis Type I; Tuberous Sclerosis Complex
Keywords: Von Recklinghausen's disease; Bourneville's disease; Cognitive variability; Loss of heterozygosity
MeSH Terms: conditions — Neurofibromatosis 1; Tuberous Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neurofibromatosis type I (NF1): Monozygotic twin pairs with genetically confirmed Neurofibromatosis type I
- Tuberous Sclerosis Complex (TSC): Monozygotic twin pairs with genetically confirmed Tuberous Sclerosis Complex

SUMMARY:
Both Neurofibromatosis type 1 (NF1) and Tuberous Sclerosis Complex (TSC) are highly heterogeneous diseases. Cognitive features seem to vary widely even between family members carrying the same mutation. This phenotypic variability is not well understood, but is generally assumed to be caused by modifier genes which regulate the affected pathways. However, recent studies brought forward an alternative explanation for the phenotypic variability. Post-mortem studies showed that second hit mutations causing loss of the second ('healthy') allele are more widespread than previously believed. These loss of heterozygosity (LOH) mutations cause bi-allelic loss of the disease-linked gene and are known to cause the gross of somatic features in both diseases (like neurofibromas and hamartomas). Hence, it could be the stochastic occurrence of second-hit mutations in the brain are the cause of the variable cognitive phenotypes.

To investigate to what extent these LOH mutations in the brain contribute to the phenotype and to what extent this variation is due to genetic modifiers factors is unknown. The investigators therefore propose to elucidate this variability by comparing the correlation of cognitive features of monozygotic twins with NF1 or TSC to healthy twins in the population. If modifier genes are the cause of the variability of cognitive features in NF1 and TSC the investigators expect that the variability in cognitive tests in monozygotic twins is the same as monozygotic twins in the healthy population. However, if the variability is caused by the occurrence of LOH mutations, the investigators expect to have a lower correlation in our monozygotic patients compared to the healthy twins.

ELIGIBILITY:
Inclusion Criteria:

* The participant is part of a monozygotic twin pair (which is genetically confirmed);
* NF1 or TSC patients with a genetically confirmed diagnosis;
* Oral and written informed consent by participant in case ≥ 18 years of age.
* Oral and written informed consent by both caregivers and assent by participant in case of minor participants.

Exclusion Criteria:

* A potential subject of whom the twin sibling is not willing or able to participate in this study, will be excluded from participation in this study.
* Symptomatic brain pathology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Monozygotic twin pairs with genetically confirmed Neurofibromatosis type I or Tuberous Sclerosis Complex
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of full intelligence quotient | 1 day
  Depending on age and cognitive development: Bayley Scales of Infant Development (BSID-III) or Wechsler Scale of Intelligence (Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III) or Wechsler Intelligence Scale for Children (WISC-III) or Wechsler Adult Intelligence Scale (WAIS-III) )

SECONDARY OUTCOMES:
Correlation of word reading ability | 1 day
  One-minute word-reading test
Correlation of attention problems | 1 day
  Conners ADHD rating scale
Correlation of behavioural problems | 1 day
  Child Behaviour Checklist or Adult Behaviour Checklist (CBCL/ABCL)
Correlation of autistic features | 1 day
  Social Responsiveness Scale (SRS)
Correlation of visuospatial judgement (NF1 twins only) | 1 day
  Judgement of Line Orientation (JLO)
Correlation of executive control (TSC twins only) | 1 day
  Trail-Making Test parts A & B (TMT)

CONTACTS AND LOCATIONS:
Overall Officials: Ype Elgersma, Prof., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands